CLINICAL TRIAL: NCT04577053
Title: Pulsed ElectroMagnetic Field Therapy With Square Wave Forms and Artificial Intelligence Within the Software Interface for Individualised, Bespoke Bio-Electromagnetic Therapy to Treat Symptoms of Chronic Lyme Disease Remaining After Antibiotics Treatment
Brief Title: PEMF Therapy to Treat Lingering Symptoms of Lyme Disease After Treatment With Antibiotics
Acronym: PEMF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It was discovered during the study that Lyme Disease is a bio warfare weapon made in USA. (See "Bitten" by Kris Newby.) The second reason for stopping the study is lack of participant responses, likely due to lack of payment for completing surveys.
Sponsor: Kasey Phifer (Other)
Responsible Party: Sponsor-Investigator, Kasey Phifer, CEO and Lead Practitioner, The National Centre for ElectroMagnetic Therapies CIC
Organization: The National Centre for ElectroMagnetic Therapies CIC (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEMF-BRI-Lyme-Disease-2020; Bioresonance Biofeedback (Other: Biofeedback Centre Bristol LTD)
Record Dates: First submitted 2020-09-17; First posted 2020-10-06 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Lyme Disease; Lyme Neuroborreliosis; Lyme Arthritis; Unknown Origin Fever
MeSH Terms: conditions — Lyme Disease; Lyme Neuroborreliosis; Fever of Unknown Origin

STUDY DESIGN:
Intervention Model Description: Control group and treatment group, no placebo
Who Masked: Outcomes Assessor
Masking Description: The independant analyst will assess the results provided in the survey, which are collected by a third party (the Google Forms app) and therefore cannot be tampered with by the Investigator. Participants complete surveys on their own mobile devices or computers at home, without any possible supervision or influence by the Investigator. The Participants are each assigned a code with which they complete the surveys on-line. The codes do not imply hierarchy (e.g. 'Alpha'), do not include numbers so as not to prime participants' answers, and have been carefully selected to remain neutral from gender, nationality, ethnicity or religious references.
  Participants have been allocated randomly using a web-based random number generator. (Screenshots of results along with participants can be requested from the Investigator.)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PEMF Therapy (Experimental): Pulsed ElectroMagnetic Field Therapy using square wave forms. In addition to set, pre-defined frequencies to aid the body's own immune system, the Artificial Intelligence incorporated into the software used will suggest a variety of frequencies to be administered during treatment. Due to the software's selection, these recommendations or selections from the software will likely be different in each treatment session.
  Interventions: Device: Scientific Consciousness Interface Operations (SCIO) Class II FDA approved medical device
- Control (No Intervention): Control group will not receive treatment.

INTERVENTIONS:
Device: Scientific Consciousness Interface Operations (SCIO) Class II FDA approved medical device — Manufactured by QX World Ltd. in Budapest, Hungary
  Other Names: INDIGO, QXCI, QUEX S, QUEX ED
  Arms: PEMF Therapy

SUMMARY:
Overview

PEMF Therapy for relief or reduction of lingering symptoms after antibiotic treatment of Lyme disease of participants in the UK.

Symptoms monitored:

Muscle ache, myalgia, muscle pain that is acutely located and/or 'wandering' (different location on different days) Aching joints Headache Fatigue, general tiredness, loss of energy, general exhaustion Mild, recurrent fever and/or chills occurring regularly Lack of oxygen in blood, feelings of 'air hunger', too high carbon dioxide levels in blood

DETAILED DESCRIPTION:
Hypothesis Period measured and observed: 18 months (Includes before treatment, during the 4-8 weeks of treatment and post treatment)

Control Group Control Group symptoms will remain the same or increase (deteriorate or worsen) by 10-20% over the period observed.

The Control Group is not asked to nor required to abstain from any other forms of treatment during the 10 month observational period; Persons in the Control Group are free to - but not encouraged to - pursue holistic, complementary and mainstream medicine for their symptoms related to contraction of Lyme Disease and any other illness that may arise.

In the event of receiving treatment or taking medicine, this information is to be passed along for data collection in the regular surveys. This will be taken into consideration when evaluating the results of the trial and hypothesis.

Test Group Test Group symptoms will improve (be reduced or eliminated) by 50-75% over the period observed; In particular, the largest improvement will be achieved during the 8 weeks of treatment. After treatment, there may be a slight improvement of symptoms, however, the improvement achieved during treatment is expected to remain the same over the next 7.5 months following treatment with the exception of re-infection or contraction of a different disease or illness.

The Test Group is not asked to nor required to abstain from any other forms of treatment during the 10 month observational period; Persons in the Control Group are free to - but not encouraged to - pursue holistic, complementary and mainstream medicine for their symptoms related to contraction of Lyme Disease and any other illness that may arise.

In the event of receiving treatment or taking medicine, this information is to be passed along for data collection in the regular surveys. This will be taken into consideration when evaluating the results of the trial and hypothesis.

Measurement (What the Investigator is Measuring and Observing in Response to Testing) and Weighting

Measurement: 1 to 100 Scale Worsening/decline or improvement/reduction of symptoms will be measured by the information collected in the surveys. Answers to questions are given subjectively by the participants themselves on a scale of 1 to 100, with 1 being the worst possible or imaginable and 100 being the best possible or imaginable. For example, the worst imaginable answer of "1" to the question of mobility/movement would be in the event that the participant is in a wheelchair or coma. Being confined to a wheelchair is certainly more mobile than lying in a comatose state, however, the answers to each question are subjective and so the participant might believe that a wheelchair would be the worst measure of mobility for him or her.

Weighting of Answers To weight the improvement or decline respectively for each participant, the average of the first three and last three surveys will be taken. This is to rule out any possible statistical outliers or anomalies due to the participant possibly having a 'bad day' or coincidental other illness such as a head cold.

Example Question:

Rate overall energy level on a scale of 1 to 100, where 1 is the lowest imaginable and 100 is the best, pre-Lyme Disease level possible.

Example Answers:

Participant A First survey: 45 Second survey: 40 Third survey: 48 25th survey (third to last): 80 26th survey (second to last): 83 27th survey (last or final): 80

Weighting here would be calculated in the following way:

Starting point or "zero point" is the average of the first three surveys

* ( 45 + 40 + 48 ) / 3 = 44.33 Ending point is the average of the last three surveys
* ( 80 + 83 + 80 ) / 3 = 81 An improvement of 100% for this participant would be from 44.33 at the starting point up to 100 at the ending point, what is to be considered a full recovery or full elimination of symptoms. The breadth of full recovery therefore contains a different amount of scala numbers for each participant, because a full recovery is based individually on each participant. This is to avoid an increase or decrease of more than 100%.

Using this example:

No improvement would be from 44.33 to [44-44.49], an increase of approximately 0 = 0% Full recovery would be from 44.33 to 100, an increase of 55.67 = 100% Amount of improvement in the example is from 44.33 to 81, an increase of 36.67; It is then calculated 36.67 / 55.67 = 68.9%

Participant B (Example Answers) First survey: 30 Second survey: 25 Third survey: 25 25th survey (third to last): 80 26th survey (second to last): 83 27th survey (last or final): 80

Weighting here would be calculated in the following way:

Starting point or "zero point" is the average of the first three surveys

* ( 30 + 25 + 25 ) / 3 = 26.67 Ending point is the average of the last three surveys
* ( 80 + 83 + 80 ) / 3 = 81 An improvement of 100% for this participant would be from 26.67 at the starting point up to 100 at the ending point, what is to be considered a full recovery or full elimination of symptoms.

Using this example:

No improvement would be from 26.67 to [26.5-27], an increase of approximately 0 = 0% Full recovery would be from 26.67 to 100, an increase of 73.33 = 100% Amount of improvement in the example is from 26.67 to 81, an increase of 54.33; It is then calculated 54.33 / 73.33 = 74.1%

More information can be found published on the investigator's website: https://biofeedbackcentrebristol.co.uk/lyme-disease-clinical-trial/

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis from GP confirming Lyme disease and/or
* Blood test confirming Lyme disease and/or
* Symptoms that correlate to Lyme disease without diagnosis from GP. This is called "self diagnosis" and because 80% of the trial is focused on treating symptoms and not the spirochetes, bacteria or small cysts of Lyme disease, the results are expected to be largely the same

Exclusion Criteria:

* Persons currently undergoing antibiotic treatment for Lyme or other conditions
* Persons who were prescribed antibiotics but did not or could not take them

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
Overall Energy Levels | 18 months
  This is inversely describing fatigue, chronic fatigue and exhaustion which is a common symptom of Lyme Disease.
Myalgia | 18 months
  This will be described to participants in an easy-to-understand 'layman' terminology. Words here include e.g. muscle ache, soreness of muscles.
Joint stiffness | 18 months
  Stiffness, soreness and lack of range of motion in any and all joints
Depression | 18 months
  This is measuring the participant's own subjective feelings of mood and depression, not a clinical diagnosis.
Fever/Chills | 18 months
  mild, recurrent fever is a common symptom of Lyme Disease. Temperature will be measured by the participants themselves should they suffer from this.

SECONDARY OUTCOMES:
Ability to Breathe | 18 months
  'Air Hunger' or the feeling of not getting enough oxygen when breathing
Encephalitis | 18 months
  Inflammation of the brain and/or spinal cord measured using the scan built into the software to confirm whether any is present in absence of medical diagnosis. Patients will report on symptoms of encephalitis, i.e. confusion, seizures, difficulty speaking, sudden changes in behaviour
Brain Fog | 18 months
  This is most likely due to hormone imbalance which results in depression, insomnia, confusion and other symptoms.
Nerve pain / damage | 18 months
  damage to the nerves resulting in loss of fine or gross motor skills, shooting pains along nerves

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - The Bristol Centre for Biofeedback, Bristol
  - The National Centre for Electromagnetic Therapies CIC, Weston

IPD SHARING:
Plan to Share IPD: Yes
Via spreadsheet and cloud sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will remain permanently available. Only participant personal data is protected under GDPR and will need special written consent prior to sharing. Otherwise, all methodology, questions, protocol and forms are being made available online.
Access Criteria: none, no login necessary. Contact the investigator if data protected under GDPR is desired, such as participants' dates of birth, names and nationalities (countries of birth)
URL: https://ncet.co.uk/clinical-trial-lyme-disease/

DOCUMENTS (1):
  • Study Protocol (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/53/NCT04577053/Prot_000.pdf